CLINICAL TRIAL: NCT03555084
Title: Quality Control of CE-Certified Phonak Hearing Aids - 2018_07
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Sonova2018_07
Record Dates: First submitted 2018-05-07; First posted 2018-06-13 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device: Extension of Phonak Virto B-Titanium (Experimental): The extension of Phonak Virto B-Titanium will be fitted to the participants individual Hearing loss.
  Interventions: Device: Extension of Virto B-Titanium
- Device: Phonak Virto B-Titanium (Active Comparator): The Phonak Virto B-Titanium will be fitted to the participants individual Hearing loss.
  Interventions: Device: Virto B-Titanium

INTERVENTIONS:
Device: Extension of Virto B-Titanium — In ear Hearing aid device individually modeled to ear canal geometry to compensate an individual Hearing loss.
  Arms: Device: Extension of Phonak Virto B-Titanium
Device: Virto B-Titanium — In ear Hearing aid device individually modeled to ear canal geometry to compensate an individual Hearing loss.
  Arms: Device: Phonak Virto B-Titanium

SUMMARY:
Phonak Hearing Systems pass through different development and study stages. At an early stage, feasibility studies are conducted to investigate new algorithms, features and functions in an isolated manner. If the benefit is proven, their performance is then investigated regarding interdependency between all available algorithms, features and functions running in parallel in a hearing aid (pivotal/pre-validation studies) and, as a result, they get optimized. Afterwards, and prior to product launch, the Phonak Hearing Systems undergo a final quality control in terms of clinical trials. This is a pre-validation study, investigating optimized algorithms, features, functions and wearing comfort. This will be a clinical evaluation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* Adult hearing impaired persons (minimum age: 18 years) with or without experience with hearing aids
* Good written and spoken (Swiss) German language skills
* Healthy outer ear
* Ability to fill in a questionnaire (p/eCRF) conscientiously
* willingness to wear custom made Hearing aids
* Informed Consent as documented by signature
* Benefit with TFG tool at least on one ear

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments in Stäfa (Switzerland)
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* Inability to produce a reliable hearing test result
* Limited dexterity (not able to change a 10size Hearing aid battery)
* no Benefit of the TFG tool on both ears
* Known psychological problems
* Central hearing disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

PRIMARY OUTCOMES:
Visibility and Wearing Comfort | 3 weeks
  The primary objective of this study is to evaluate if Virto B-Titanium hearing aids measured with the Titanium FitGuide (TFG) (extension of Virto B-Titanium) are less visible (deeper) than modeling without TFG (Virto B-Titanium) while maintaining wearing comfort on adult participants (new and existing users) with mild to moderately-severe hearing loss (M and P receiver ).

SECONDARY OUTCOMES:
Measurement of acoustic Feedback Thresholds | 3 weeks
  Secondary objective is to compare the acoustic feedback thresholds of the TFG- and without TFG- modeled devices in regard of an adequate sealing effect of the respective devices. Thereby, feedback thresholds, measured with the Phonak Target fitting software, must be comparable to average feedback threshold values of the respective shell forms (IIC / CIC). Acceptable feedback thresholds must guarantee an insertion gain [in dB SPL] of at least 20 dB in a specific frequency range.

OTHER OUTCOMES:
TFG Fitrate | 3 weeks
  Another objective is to investigate whether at least 50% of the screened population will get a deeper fitted device by the use of the TFG tool, proven by modelling software

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Canton of Zurich, Switzerland